CLINICAL TRIAL: NCT02463591
Title: Reversal of Anticoagulant Effect of Dabigatran® by Prothrombin Complex Concentrate (Beriplex®), Assessed With a Novel Method of Blood Loss Measurement
Brief Title: Reversal of Dabigatran With Prothrombin Complex Concentrate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Boehringer Ingelheim (Industry); CSL Behring (Industry)
Responsible Party: Principal Investigator, Pieter W. Kamphuisen, MD PhD, Prof. dr., University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BI 1160.203; 2014-002204-24 (EudraCT Number)
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Drug Action Reversal
Keywords: Direct Thrombin Inhibitor; Prothrombin Complex Concentrate; Dabigatran Etexilate; Beriplex; Shed Blood; Washed Blood; Fibrinopeptide A
MeSH Terms: conditions — Hemophilia B | interventions — factor IX, factor VII, factor X, prothrombin drug combination; Factor IX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beriplex 50 IU/Kg (Experimental): Cross over design: After therapy with Dabigatran Etexilate 300mg BID for 2.5 days, subjects will receive a single dose of Beriplex 50 IU/Kg. After a 10 day minimum wash-out period subjects will receive the alternative treatment (Placebo).
  Interventions: Drug: Beriplex
- Placebo (Placebo Comparator): Cross over design: After therapy with Dabigatran Etexilate 300mg BID for 2.5 days, subjects will receive a single dose of Placebo identically in appearance to Beriplex 50 IU/Kg. After a 10 day minimum wash-out period subjects will receive the alternative treatment (Beriplex).
  Interventions: Drug: Beriplex

INTERVENTIONS:
Drug: Beriplex — Beriplex 50 IU/Kg i.v. , single dose.
  Other Names: Prothrombin Complex Concentrate; RVG 101094; B02BD01

SUMMARY:
The purpose of this study is to investigate whether Prothrombin Complex Concentrate (PCC) is effective in reversing the anticoagulant effect of Dabigatran, as assessed by two modified skin-bleeding tests.

DETAILED DESCRIPTION:
There is currently no treatment widely available for immediate reversal of Dabigatran anticoagulant effects, e.g. in case of major bleeding or when emergency surgery or invasive procedures are indicated.

Treatment with prothrombin complex concentrate (PCC) seems effective in reducing blood loss in animal models, but previous studies in humans have failed to show an effect on blood coagulation parameters. Recently, two novel methods of skin blood loss, one called "shed blood" and another "washed blood" were able to measure effects of anticoagulation, either as the inhibition of fibrin formation at the wound site by measuring Fibrinopeptide A (FPA) or as elevated blood loss, respectively, after oral administration of Dabigatran in healthy volunteers.

The investigators hypothesise that the shed/washed blood methods are able to measure Dabigatran reversal following administration of PCC (Beriplex).

The study will be performed as a randomised double blind cross-over study and 12 healthy human male subjects will be enrolled. Subjects will take Dabigatran 300 mg b.i.d. on day -2, -1 and 0. After the fifth dose (on day 0), subjects will be randomised to receive Beriplex (50 IU/kg) or a similar volume of saline as a single bolus dose i.v. over 20 minutes. After a 10 day minimum wash-out period this procedure will be repeated, and the alternative treatment (Saline or Beriplex) is administered.

The Shed / Washed Blood measurements will be performed at different time points before and after starting oral anticoagulants and before and after administration of Beriplex/Saline.

In addition to the Shed / Washed blood tests, several ex vivo standard coagulation tests will be performed. These include: activated partial thromboplastin time (aPTT), prothrombin time (PT), diluted thrombin time (DTT/Hemoclot), Dabigatran plasma levels (using liquid chromatography-tandem mass spectrometry (LC-MS/MS)), endogenous thrombin generation (ETG) and pre and post factor II, VII, IX and X.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age between 18 and 50 years
* Weight <100 kg
* Signed informed consent
* eGFR ≥ 80ml/min*1.73m2

Exclusion Criteria:

* History of allergic reaction to blood products
* Current participation in any other investigational drug study or within the past 30 days
* Increased bleeding tendency or history of thrombosis
* Anticoagulant medication, platelet aggregation inhibitors or NSAIDs
* Use of any medication 14 days before start of dabigatran intake

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Inhibition of the anticoagulant effect of Dabigatran, assessed by the "shed and washed blood" methods | Before Dabigatran (Baseline, T= day-2), After Dabigatran / Before PCC (T= day 0), After Dabigatran / After PCC (T=40 min.), After Dabigatran / After PCC (T=360 min.)
  The Shed blood test allows assessment of thrombin activity and subsequent fibrinogen conversion to fibrin in vivo by measuring fibrinopeptide A (FPA) generation. A standardized wound, using a disposable device (Surgicutt® Adult) is made on the volar surface of the forearm, from which blood is collected during 4 minutes. The total amount of shed blood is measured in addition to Fibrinopeptide A levels. FPA levels are compared to FPA levels in systemic venous samples collected at corresponding timepoints.
  The washed blood test measures both the time until bleeding stops and sensitively measures small volumes of blood loss as area under the curve (AUC).

SECONDARY OUTCOMES:
Change in Standard Coagulation Assays before / after Dabigatran and before / after PCC. | Before Dabigatran (Baseline, T= day-2), After Dabigatran / Before PCC (T= day 0), After Dabigatran / After PCC (T=20 min., T=40 min., T=60 min., T=120 min., T=240 min., T=360 min.
  aPTT, PT, Diluted Thrombin Time (Hemoclot), Dabigatran Plasma Levels, Endogenous thrombin generation, pre- and Post coagulation factor II / VII / IX / X

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Willem Kamphuisen, Prof. Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolzt M, Eder M, Weltermann A, Entlicher J, Eichler HG, Kyrle PA. Comparison of the effects of different low molecular weight heparins on the hemostatic system activation in vivo in man. Thromb Haemost. 1997 Aug;78(2):876-9. PMID 9268188